CLINICAL TRIAL: NCT02140034
Title: Extensive Peritoneal Lavage After Curative Gastrectomy for Gastric Cancer: A Randomised Controlled Trial (EPL Study)
Brief Title: Extensive Peritoneal Lavage After Curative Gastrectomy for Gastric Cancer: A Randomised Controlled Trial
Acronym: EPL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPL Study; 2013/00172 (Other: DSRB)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Gastric Cancer
Keywords: Extensive Peritoneal Lavage; Overall Survival; Disease Free Survival; Peritoneal Recurrence Rate; T3 and T4 Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Arm: Extensive Peritoneal Lavage (Experimental): The peritoneal cavity of subject will be washed with 10 liters of warmed normal saline (1 liter per cycle for 10 cycles) . The abdomen will be closed as per standard
  Interventions: Procedure: Extensive Peritoneal Lavage
- Control Arm: Standard Treatment (No Intervention): The peritoneal cavity of subjects will be washed with 2 liters or less of warmed normal saline. The abdomen will be closed as per standard.

INTERVENTIONS:
Procedure: Extensive Peritoneal Lavage
  Arms: Study Arm: Extensive Peritoneal Lavage

SUMMARY:
This study is carried out to determine the merit and reliability of extensive intraoperative peritoneal lavage as a preventive strategy

Hypothesis: EPL significantly improve the overall survival of patients by reducing the risk of peritoneal recurrence

DETAILED DESCRIPTION:
Gastric cancer is the second most common cause of cancer death worldwide. Surgery is the mainstay treatment for cure. Peritoneum is a common site of recurrence and the prognosis in patients with peritoneal recurrence is dismal. Hence, prevention is essential to patient's outcomes. In patients with serosal invasion, about half experience peritoneal recurrence within first 2 years after surgery, even after curative surgery. Peritoneal metastasis is caused by the implantation of free cancer cells in the peritoneal cavity exfoliated from the primary tumor before or during curative surgery. It is well known that cancer cells spillage could occur during surgery due to manipulation or even after lymph node dissection. If we can remove these free exfoliated cancer cells on the peritoneal lining, we may reduce the risk of tumor recurrence.

Recently, a study has demonstrated a dramatic reduction of peritoneal recurrence with extensive peritoneal lavage (EPL) in patients who underwent curative resection of gastric cancer. EPL was performed after the curative operation . The peritoneal cavity was washed with normal saline which is then followed by the complete aspiration of the fluid. This procedure was done 10 times using 1 liter of normal saline. The method was based on the 'limiting dilution theory' in which the method can dilute the number of free cancer cells to minimal hence reduce the risk of tumor implantation. In this study, among patients with microscopic peritoneal metastasis, peritoneal recurrence developed in 40% of patients with EPL and surgery, compared to 89.7% in patients with surgery alone. EPL carries minimal risk to patients. It is simple and inexpensive, and it is not time consuming. Hence, it may be an effective strategy for treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have T3 (subserosal) or T4 (serosal) disease based on CT scan and intra-operative inspection with any N staging and M0 gastric cancer.
* Patients planned for open or laparoscopic gastrectomy.
* Patients undergoing gastrectomy with curative intent.
* Lower age limit of research subjects 21 years old and upper age limit of 80 years old.
* Ability to provide informed consent

Exclusion Criteria:

* Patients who undergo a palliative gastrectomy.
* Patients who undergo a gastrectomy as emergency.
* Vulnerable persons under age of 21.
* Patients receiving neoadjuvant therapy.
* Patients presented with life-threatening bleeding from tumour
* ASA score of 4 & 5
* Patients with another primary cancer within last 5 years
* Patients with gross peritoneal and liver metastasis at surgery.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years

SECONDARY OUTCOMES:
Disease Free Survival | 3 years
Peritoneal Recurrence Rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy So, MBChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Misawa K, Mochizuki Y, Ohashi N, Matsui T, Nakayama H, Tsuboi K, Sakai M, Ito S, Morita S, Kodera Y. A randomized phase III trial exploring the prognostic value of extensive intraoperative peritoneal lavage in addition to standard treatment for resectable advanced gastric cancer: CCOG 1102 study. Jpn J Clin Oncol. 2014 Jan;44(1):101-3. doi: 10.1093/jjco/hyt157. Epub 2013 Nov 27. PMID 24287077
- [Background] Kuramoto M, Shimada S, Ikeshima S, Matsuo A, Yagi Y, Matsuda M, Yonemura Y, Baba H. Extensive intraoperative peritoneal lavage as a standard prophylactic strategy for peritoneal recurrence in patients with gastric carcinoma. Ann Surg. 2009 Aug;250(2):242-6. doi: 10.1097/SLA.0b013e3181b0c80e. PMID 19638909
- [Derived] Yang HK, Ji J, Han SU, Terashima M, Li G, Kim HH, Law S, Shabbir A, Song KY, Hyung WJ, Kosai NR, Kono K, Misawa K, Yabusaki H, Kinoshita T, Lau PC, Kim YW, Rao JR, Ng E, Yamada T, Yoshida K, Park DJ, Tai BC, So JBY; EXPEL study group. Extensive peritoneal lavage with saline after curative gastrectomy for gastric cancer (EXPEL): a multicentre randomised controlled trial. Lancet Gastroenterol Hepatol. 2021 Feb;6(2):120-127. doi: 10.1016/S2468-1253(20)30315-0. Epub 2020 Nov 27. PMID 33253659